CLINICAL TRIAL: NCT04788225
Title: Assessment of Balance and Function After Lateral Ankle Ligament Repair
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, İnci Hazal Ayas, Principal Investigator, Gazi University
Other Study IDs: IAyas
Record Dates: First submitted 2021-02-27; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Complete Tear, Ankle, Lateral Ligament; Postural Balance; Physical Functional Performance
Keywords: Lateral ankle ligaments repair; Postural Balance; Physical Functional Performance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with ATFL repair by arthroscopic method: Patients who have passed at least 1 year after the operation Unilateral arthroscopic ATFL repair Between the ages of 18-65 Volunteer to participate in the study Without any orthopedic conditions, neuromuscular disease, balance disorder, cognitive disorder No history of fracture and surgical operation of the lower extremity
  Interventions: Other: Balance assessment; Other: Functionality assessment; Other: Performance assessment; Other: ROM assessment
- Control group: Between the ages of 18-65 Volunteer to participate in the study Healthy individuals with no disease
  Interventions: Other: Balance assessment; Other: Functionality assessment; Other: Performance assessment; Other: ROM assessment

INTERVENTIONS:
Other: Balance assessment — Static balances will be measured with the Biodex-BioSway 950-462 static balance device according to 3 different standard test procedures (Postural Stability Test, Stability Limit Test and Modified Sensori Organization Test) in single foot stance and double foot stance.
  Dynamic balances will be evaluated with the Y balance test.
  Other Names: Clinical assessment
Other: Functionality assessment — Functionality will be evaluated with the Lower Extremity Functional Scale and AOFAS (American Orthopedic Foot and Ankle Society Ankle-Hindfoot Scale)
  Other Names: Clinical assessment
Other: Performance assessment — Performance evaluation will be made with a single leg jump test and time up and go test.
  Other Names: Clinical assessment
Other: ROM assessment — Range of motion (ROM) of the ankle will be measured with an electrogonyometer in dorsi-plantar flexion.
  Other Names: Clinical assessment

SUMMARY:
Approximately 85% of ankle injuries are lateral region injuries.Surgical repair of lateral ligaments is indicated if there is more than 20 degrees of varus or more than 15 mm translation, if conservative treatment is ineffective and degree of damage is high and chronic instability has developed.After the surgery in addition to pain and edema control, weight transfer is not performed on the ankle for 6 weeks.Therefore, this process may adversely affect the muscle strength and range of motion of the ankle, and lower extremity performance and muscular synergies of balance.Although pathological changes caused by ligament damage have been investigated very well in the literature, it is not clear how surgical repair affects these changes. In our study we aim to investigate post-surgical changes.

Primary aim of the study is to evaluate the balance parameters of individuals who have undergone anterior talofibular ligament and / or calcaneofibular ligament repair, and its secondary purpose is to evaluate lower extremity performance, ankle functionality, pain, range of motion and muscle strength and compare them with healthy individuals.

Our hypothesis is that the balance, lower extremity performance and functionality, pain, range of motion and muscle strength of patients who have undergone ankle lateral ligament repair are worse than healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have passed at least 1 year after the operation Unilateral arthroscopic ATFL repair Volunteer to participate in the study

Exclusion Criteria:

* Any orthopedic conditions, neuromuscular disease, balance disorder, cognitive disorder, history of fracture and surgical operation of the lower extremity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone ATFL repair surgery at Gazi University Hospital The healthy control group will consist of patient relatives or volunteers to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-02-12 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Static balance assessment-Postural Stability Test | 1 year postoperatively
  Postural Stability will be measured with the Biodex-BioSway 950-462 static balance device in single foot stance and double foot stance.
Static balance assessment-Stability Limit Test | 1 year postoperatively
  Stability Limit will be measured with the Biodex-BioSway 950-462 static balance device in double foot stance.
Static balance assessment-Modified Sensori Organization Test | 1 year postoperatively
  Modified Sensori Organization will be measured with the Biodex-BioSway 950-462 static balance device in double foot stance.
Dynamic balance assessment | 1 year postoperatively
  Dynamic balances will be evaluated with the Y balance test.

SECONDARY OUTCOMES:
Jumping performance assessment | 1 year postoperatively
  Performance evaluation will be made with a single leg jump test.
Walking ability | 1 year postoperatively
  Performance evaluation will be made with time up and go test.
Lower limb functionality assessment | 1 year postoperatively
  Functionality will be evaluated with the Lower Extremity Functional Scale.
Foot and ankle functionality assessment | 1 year postoperatively
  Functionality will be evaluated with the AOFAS (American Orthopedic Foot and Ankle Society Ankle-Hindfoot Scale)
ROM assessment | 1 year postoperatively
  Range of motion (ROM) of the ankle will be measured with an electrogonyometer in dorsi-plantar flexion.

CONTACTS AND LOCATIONS:
Overall Officials: seyit çıtaker, Study Director — Gazi University
Locations (1):
- Inci Ayas, Ankara, Turkey (Türkiye)